CLINICAL TRIAL: NCT00157703
Title: A Staged Phase 1 Study of the Treatment of Malignant Glioma With G207, a Genetically Engineered HSV-1, Followed by Radiation Therapy
Brief Title: G207 Followed by Radiation Therapy in Malignant Glioma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MediGene (Industry)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Alice Chen, MediGene
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT2001
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2008-12-16 (Estimated); Status verified 2008-12

CONDITIONS: Malignant Glioma
Keywords: Malignant glioma; Glioblastoma multiforme; GBM; Gliosarcoma; Anaplastic astrocytoma; Brain cancer; Brain tumor; Glioma; recurrent/progressive malignant glioma
MeSH Terms: conditions — Glioma; Glioblastoma; Gliosarcoma; Astrocytoma; Brain Neoplasms; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: G207 — 1 x 10E9 plaque forming units, administered by stereotactic injections into the tumor (single administration)

SUMMARY:
This is an open-label, single site study to evaluate the safety and tolerability of intratumoral administration of G207 followed by treatment with radiation therapy in patients with recurrent/progressive malignant glioma.

This study is a two stage phase 1 study, in which a de-escalating dosing scheme will be used, i.e. the first patients will receive the higher dose and if excessive toxicity occurs, the dose will be reduced for the following patients. The purpose of the dose de-escalation phase is to find the best safe dose of G207.

In the first stage of the study, treatment with G207 will be followed by focal radiation therapy on the following day, and in the second stage treatment with G207 will be followed by gamma knife surgery also on the following day.

All patients will return to the clinic 28 days and 3, 6, 9 and 12 months after G207 administration at which time clinical assessments will be performed, and will be followed for safety and survival at clinic visits or by telephone every 3 months for up to 2 additional years and annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically proven residual/recurrent glioblastoma multiforme, gliosarcoma or anaplastic astrocytoma which is progressive despite radiotherapy or chemotherapy
2. Failed external beam radiotherapy > 5,000 CGy at least 4 weeks prior to enrollment
3. Residual/recurrent lesion must be ≥ 1.0 cm and (for Stage 2 only) ≤ 4 cm in diameter as determined by magnetic resonance imaging (MRI)
4. Normal hematological, renal and liver function

   * Absolute neutrophil count > 1500/mm3
   * Platelets > 100,000/mm3
   * Prothrombin time (PT) or partial thromboplastin time (PTT) < 1.3 x control
   * Creatinine < 1.7 mg/dl
   * Total bilirubin < 1.5 mg/dl
   * Transaminases < 4 times above the upper limits of the institutional norm
5. Karnofsky Performance Status score ≥ 70
6. Age > 19 years-old
7. Capable of giving informed consent
8. Must be willing to practice an effective barrier method of birth control for 2 months post G207 inoculation, whether male or female
9. Females of childbearing potential: negative pregnancy test within 24 hours prior to G207 administration

Exclusion Criteria:

1. Surgical resection within 4 weeks of enrolment
2. Acute infection, granulocytopenia or medical condition precluding surgery
3. Pregnant or lactating females
4. History of encephalitis, multiple sclerosis, or other central nervous system (CNS) infection
5. Tumor involvement which would require ventricular, brainstem, basal ganglia, or posterior fossa inoculation or would require access through a ventricle in order to deliver treatment or tumor involving both hemispheres or with subependymal/cerebral spinal fluid (CSF) dissemination
6. Tumor position that could, in the Investigator's opinion, pose the risk of penetration of the cerebral ventricular system during inoculation with the study drug (Note: If penetration of the ventricular system is suspected or confirmed, G207 administration must be aborted.)
7. Tumor locations that would expose the patient to unacceptable risk with radiation therapy
8. Prior participant in experimental viral therapy (e.g., adenovirus, retrovirus or herpesvirus protocol)
9. Prior participant in chemotherapy, cytotoxic therapy, immunotherapy or gene therapy protocol within 6 weeks of enrolment
10. Required steroid increase within 2 weeks prior to injection
11. HIV seropositive
12. Concurrent therapy with any drug active against herpes simplex virus (HSV) (acyclovir, valaciclovir, penciclovir, famciclovir, ganciclovir, foscavir, cidofovir)
13. Active oral or genital herpes lesion
14. Any contraindication for undergoing MRI such as pacemakers, infusion pumps, ferromagnetic aneurysm clips, metal prostheses, etc.
15. Radiation treatment volume of greater than 4 cm maximum diameter (Stage 2 only)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2005-05; Primary Completion 2008-10 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Adverse events | from 1st dose to end of study visit

SECONDARY OUTCOMES:
Radiographic response | Withdrawal or death of last patient
Performance scale | Last patient out
Overall survival | Withdrawal or death of last patient
Immune response | Last patient out
Presence of G207 in blood and saliva | Last patient out

CONTACTS AND LOCATIONS:
Overall Officials: Axel Mescheder, M.D., Study Director — Medigene AG
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

REFERENCES:
- [Derived] Markert JM, Razdan SN, Kuo HC, Cantor A, Knoll A, Karrasch M, Nabors LB, Markiewicz M, Agee BS, Coleman JM, Lakeman AD, Palmer CA, Parker JN, Whitley RJ, Weichselbaum RR, Fiveash JB, Gillespie GY. A phase 1 trial of oncolytic HSV-1, G207, given in combination with radiation for recurrent GBM demonstrates safety and radiographic responses. Mol Ther. 2014 May;22(5):1048-55. doi: 10.1038/mt.2014.22. Epub 2014 Feb 27. PMID 24572293